CLINICAL TRIAL: NCT05530460
Title: Comparative Study of High Performance Low-Cost Optical Coherence Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00111488; R01AG072732 (NIH)
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Optical Coherence Tomography of Retina

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OCT Imaging (Experimental)
  Interventions: Device: retinal imaging with low-cost OCT device; Device: retinal imaging with commercial OCT device

INTERVENTIONS:
Device: retinal imaging with low-cost OCT device — Retinal imaging with low-cost OCT device
Device: retinal imaging with commercial OCT device — retinal imaging with commercial OCT device

SUMMARY:
The purpose of this study is to complete performance testing of our custom optical coherence tomography (OCT) device to verify it can deliver retinal images of similar quality to a commercial OCT device.

DETAILED DESCRIPTION:
There is some evidence that certain changes in retinal structures could be an indicator of Alzheimer's disease (AD). We are developing a new technology that combines optical coherence tomography (OCT) and angle-resolved low coherence interferometry (a/LCI) to make light scattering measurements of retinal tissue structure. The objective of this device feasibility study is to compare performance characteristics of our custom OCT instrument to a commercial OCT instrument. Once we have optimized our device, we may use it in future studies to identify retinal structure changes that could be possible AD biomarkers.

For this study, the team will recruit healthy volunteers to attend one study visit that is about 30 minutes long. This visit will include examination with our custom OCT instrument, followed by examination with a commercial OCT system.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent

Exclusion Criteria:

* potentially confounding ocular conditions, such as: glaucoma, current corneal injury, retinal damage, diabetes, corrected distance visual acuity worse than 20/40
* eyes that have had intraocular surgery, other than cataract surgery

If two eyes satisfy the inclusion / exclusion criteria, both eyes will be included in the study. If only one eye satisfies the criteria, only the qualifying eye will be included in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Acceptable OCT Image Quality as Measured by Low-Cost OCT Device | during study procedures (30 minutes)
  measured by: ability to see clearly defined and recognizable structures of the retina with the low-cost OCT device.

SECONDARY OUTCOMES:
Contrast-to-Noise Ratio (CNR) | during study procedures (30 minutes)
  Measure of OCT image quality comparing level of image contrast to level of background noise. CNR = (mean of signal of region of interest [i.e., retina] - mean of background noise) divided by square root of (the square of the standard deviation of the region of interest + the square of the standard deviation of the background noise). Therefore, CNR is unitless.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wax, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No